CLINICAL TRIAL: NCT02365519
Title: A Randomized, Double-masked, Vehicle-controlled Study of LME636 in the Relief of Persistent Ocular Discomfort in Subjects With Severe Dry Eye Disease
Brief Title: LME636 in the Relief of Persistent Ocular Discomfort in Subjects With Severe Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon, a Novartis Company (Industry)
Collaborators: Novartis Institutes for BioMedical Research (Other)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LME636-2202
Record Dates: First submitted 2015-02-13; First posted 2015-02-19 (Estimated); Results first posted 2017-11-24 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-10

CONDITIONS: Dry Eye
Keywords: LME636; dry eye disease; efficacy; ocular discomfort
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LME636 (Experimental): LME636 ophthalmic solution, 1 drop (approx. 40 µL; 2.4 mg) administered topically in each eye 3 times a day (TID) for 6 weeks
  Interventions: Biological: LME636 ophthalmic solution
- Vehicle (Placebo Comparator): LME636 Vehicle, 1 drop administered topically in each eye TID for 6 weeks
  Interventions: Biological: LME636 Vehicle

INTERVENTIONS:
Biological: LME636 ophthalmic solution
  Arms: LME636
Biological: LME636 Vehicle — Inactive ingredients used as a placebo comparator
  Arms: Vehicle

SUMMARY:
The purpose of this study is to evaluate the efficacy of LME636 compared to vehicle in the reduction of ocular symptoms and to evaluate the safety and tolerability of LME636, when administered topically for up to 42 days, in subjects with severe dry eye disease.

DETAILED DESCRIPTION:
This study is organized into 2 phases. Following a 2-week identification phase, eligible subjects with severe dry eye disease (DED) will be randomized into the treatment phase and will be dispensed study treatment for 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Must sign written informed consent.
* Physician diagnosis of DED of at least 6 months prior to Visit 1.
* Must use artificial tears, gels, lubricants or re-wetting drops on a regular basis.
* Respond as "often" or "constantly" to the question "How often do your eyes feel uncomfortable?".
* Best Corrected Visual Acuity (BCVA) of 55 or greater in each eye as measured by ETDRS at Visit 1.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Presence of any acute infection or non-infectious ocular condition in either eye within 1 month of Visit 1.
* Contact lens wearers, defined as individuals who cannot be without their contact lenses for the entire duration of the study.
* Any chronic ocular degenerative condition that in the opinion of the Investigator could possibly advance during the time course of the study.
* Use of biologics treatments, such as systemic biologic anti-cytokines, including anti-TNFα drugs, or immunosuppressive therapy for the treatment of severe systemic autoimmune disorders.
* Diseases or conditions affecting the ocular surface that are associated with clinically significant scarring and or destruction of conjunctiva and/or cornea.
* Unwilling to abstain from topical ocular non-prescription medications during the course of the study, including concomitant use of artificial tears, gels, lubricants, re-wetting drops, allergy drops, etc. after Visit 2.
* Use of nasal, inhaled, systemic (including injections), or topical corticosteroids within 30 days of Visit 1.
* Women of child-bearing potential unwilling to use effective contraception methods as defined in the protocol.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2015-03-09 (Actual); Primary Completion 2015-10-16 (Actual); Study Completion 2015-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Clinical Manager, GCRA, Study Director — Alcon, A Novartis Division

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 31 investigational sites located in the US.
Pre-assignment Details: Of the 514 enrolled, 213 subjects entered the vehicle run-in period and 134 entered the randomized treatment period.
Groups:
- Vehicle Run-In: All subjects exposed to LME636 Vehicle prior to the initiation of randomized study treatment
- LME636: All subjects exposed to LME636 ophthalmic solution during randomized study treatment
- Vehicle: All subjects exposed to LME636 Vehicle during randomized study treatment
Period: Vehicle Run-In
Arm/Group | Vehicle Run-In | LME636 | Vehicle
Started | 213 | 0 | 0
Completed | 134 | 0 | 0
Not Completed | 79 | 0 | 0
Period: Randomized and Treated
Arm/Group | Vehicle Run-In | LME636 | Vehicle
Started | 0 | 69 | 65
Completed | 0 | 67 | 64
Not Completed | 0 | 2 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized and treated subjects.
Groups:
- LME636: All subjects randomized and treated with LME636 ophthalmic solution
- Vehicle: All subjects randomized and treated with LME636 Vehicle
- Total: Total of all reporting groups
Arm/Group | LME636 | Vehicle | Total
Number analyzed (Participants) | 69 | 65 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (13.05) | 58.8 (14.48) | 60.3 (13.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 54 | 115
  Male | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Global Ocular Discomfort Score at Day 71
Description: Discomfort frequency and severity (each graded on a separate 100-units scale) were assessed daily using a visual analog scale (VAS) displayed on a handheld digital Pad (electronic patient-reported outcome (ePRO)). Frequency score was in response to the question 'how often your eyes felt uncomfortable during the past 24 hours' ranging from 'Rarely' to 'All the time.' Severity score was in response to the question 'how uncomfortable your eyes felt during the past 24 hours' ranging from 'Very mildly uncomfortable' to 'Very severely uncomfortable.' The Global Ocular Discomfort Score, ranging from 0 to 100, was calculated for any given day, as the square root of the product of the discomfort frequency score multiplied by the discomfort severity score. Improvement results in a reduction of the discomfort frequency or severity, or both, translating into a reduction of the resulting Global Ocular Discomfort score as compared to baseline. A negative change from baseline indicates improvement.
Time Frame: Baseline (Day 43), Day 71
Population: This analysis population includes all randomized subjects with at least a post-baseline primary endpoint assessment excluding all subjects who met the critical deviation criteria (Per-Protocol Set). Number Analyzed is the number of subjects with data at visit.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- LME636: LME636 ophthalmic solution, 1 drop (approx. 40 µL; 2.4 mg) administered topically in each eye TID for 6 weeks
Arm/Group | LME636 | Vehicle
Number analyzed (Participants) | 67 | 64
units on a scale | -7.9 (1.45) | -3.6 (1.49)

2. Primary Outcome: Best Corrected Visual Acuity (BCVA)
Description: Visual Acuity (VA) with the subject's best spectacles or other visual corrective devices was measured using an ETDRS visual acuity chart at 3 meters (10 feet) and reported in letters read correctly. An increase (gain) in letters read indicates improvement. Both eyes contributed to the analysis.
Time Frame: Baseline (Day 43), Day 57, Day 71, Day 85
Population: This analysis population includes all subjects that received any study drug (Safety Analysis Set). Number Analyzed is the number of subjects with data at visit.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | LME636 | Vehicle
Number analyzed (Participants) | 69 | 65
letters
  Baseline (Day 43) | 80.6 (6.44) | 81.5 (5.72)
  Day 57 | 80.5 (6.82) | 81.6 (5.48)
  Day 71 | 81.6 (5.56) | 81.9 (5.89)
  Day 85: number analyzed (Participants) | 67 | 64
  Day 85 | 81.0 (5.73) | 81.6 (6.17)

3. Primary Outcome: Intraocular Pressure (IOP)
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry or Tonopen and measured in millimeters of mercury (mmHg). A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). Both eyes contributed to the analysis.
Time Frame: Baseline (Day 43), Day 57, Day 71, Day 85
Population: Safety Analysis Set. Number Analyzed is the number of subjects with data at visit.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LME636 | Vehicle
Number analyzed (Participants) | 69 | 65
mmHg
  Baseline (Day 43) | 14.8 (2.71) | 14.3 (2.63)
  Day 57 | 14.6 (2.72) | 14.1 (2.92)
  Day 71 | 14.0 (3.06) | 14.1 (2.70)
  Day 85: number analyzed (Participants) | 67 | 64
  Day 85 | 14.4 (2.68) | 14.6 (2.58)

4. Primary Outcome: Percentage of Subjects With Increase in Slit-Lamp Parameter From Baseline to Any Visit
Description: Ocular signs (cornea, lens, and iris/anterior chamber) were assessed by slit-lamp biomicroscopy. An increase indicates worsening. Only one eye contributed to the analysis.
Time Frame: Baseline (Day 43), Day 57, Day 71, Day 85
Population: Safety Analysis Set
Measure: Number; unit: percentage of subjects
Arm/Group | LME636 | Vehicle
Number analyzed (Participants) | 69 | 65
percentage of subjects
  Cornea | 0.0 | 0.0
  Lens | 0.0 | 0.0
  Iris | 0.0 | 0.0
  Anterior Chamber | 0.0 | 0.0

5. Primary Outcome: Percentage of Subjects With Increase in Dilated Fundus Parameter From Baseline to Any Visit
Description: The dilated fundus examination was performed to evaluate the health of the vitreous, retina, macula, choroid, and optic nerve. An increase indicates worsening. Only one eye contributed to the analysis.
Time Frame: Baseline (Day 43), Day 57, Day 71, Day 85
Population: Safety Analysis Set
Measure: Number; unit: percentage of subjects
Arm/Group | LME636 | Vehicle
Number analyzed (Participants) | 69 | 65
percentage of subjects
  Vitreous | 1.4 | 1.5
  Retina | 1.4 | 0.0
  Macula | 0.0 | 0.0
  Choroid | 0.0 | 0.0
  Optic Nerve | 0.0 | 0.0

6. Secondary Outcome: Percentage of Subjects With More Than 20 Units Improvement in Global Ocular Discomfort Score From Baseline at Day 71
Description: Discomfort frequency and severity (each graded on a separate 100-units scale) were assessed daily using a VAS displayed on a handheld ePRO. Frequency score was in response to the question 'how often your eyes felt uncomfortable during the past 24 hours' ranging from 'Rarely' to 'All the time.' Severity score was in response to the question 'how uncomfortable your eyes felt during the past 24 hours' ranging from 'Very mildly uncomfortable' to 'Very severely uncomfortable.' The Global Ocular Discomfort Score, ranging from 0 to 100, was calculated for any given day, as the square root of the product of the discomfort frequency score multiplied by the discomfort severity score. Improvement results in a reduction of the discomfort frequency or severity, or both, translating into a reduction of the resulting Global Ocular Discomfort score as compared to baseline.
Time Frame: Baseline (Day 43), Day 71
Population: Per-Protocol Set
Measure: Number; unit: percentage of subjects
Arm/Group | LME636 | Vehicle
Number analyzed (Participants) | 67 | 64
percentage of subjects | 17.9 | 4.7

7. Secondary Outcome: Percentage of Subjects With LME636 Serum Concentrations Below the Lower Limit of Quantification (LLOQ)
Description: Serum concentrations at each collection time point were quantitated, where possible, using a validated immunoassay method. LLOQ is defined as 0.25 ng/mL.
Time Frame: Day 15, Day 29, Day 43, Day 57, Day 71, Day 85
Population: This analysis population includes all subjects with available pharmacokinetics data (Pharmacokinetics Analysis Set).
Measure: Number; unit: percentage of subjects
Arm/Group | LME636
Number analyzed (Participants) | 69
percentage of subjects
  Day 15 | 100.0
  Day 29 | 100.0
  Day 43 (prior to administration of first dose): number analyzed (Participants) | 68
  Day 43 (prior to administration of first dose) | 98.5
  Day 57: number analyzed (Participants) | 56
  Day 57 | 82.1
  Day 71: number analyzed (Participants) | 57
  Day 71 | 71.9
  Day 85 (last day of dosing): number analyzed (Participants) | 53
  Day 85 (last day of dosing) | 67.9

8. Secondary Outcome: Percentage of Subjects With Anti-LME636 Antibodies by Visit
Description: Samples were collected and assessed for anti-LME636 antibodies.
Time Frame: Day 15, Day 29, Day 43, Day 57, Day 71, Day 85
Population: This analysis population includes all subjects with available immunogenicity data (Immunogenicity Analysis Set).
Measure: Number; unit: percentage of subjects
Groups:
- Vehicle: LME636 Vehicle, 1 drop administered topically in each eye TID for 6 weeks during randomized study treatment
- Run-In Only: LME636 Vehicle, 1 drop administered topically in each eye TID for 4 weeks with exit prior to start of randomized treatment
Arm/Group | LME636 | Vehicle | Run-In Only
Number analyzed (Participants) | 69 | 65 | 79
percentage of subjects
  Day 15: number analyzed (Participants) | 60 | 55 | 78
  Day 15 | 33.3 | 40.0 | 26.9
  Day 29: number analyzed (Participants) | 59 | 53 | 74
  Day 29 | 37.3 | 37.7 | 27.0
  Day 43 (prior to administration of first dose): number analyzed (Participants) | 69 | 63 | 63
  Day 43 (prior to administration of first dose) | 31.9 | 34.9 | 27.0
  Day 57 (Treatment Day 15): number analyzed (Participants) | 57 | 56 | 0
  Day 57 (Treatment Day 15) | 45.6 | 41.1 |
  Day 71: number analyzed (Participants) | 58 | 48 | 0
  Day 71 | 79.3 | 41.7 |
  Day 85 (last day of dosing): number analyzed (Participants) | 53 | 52 | 0
  Day 85 (last day of dosing) | 86.8 | 40.4 |

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of informed consent for the duration of a subject's participation in the study (up to 85 days).
Description: An AE was defined as any untoward medical occurrence in a subject who is administered a study treatment regardless of whether or not the event has a causal relationship with the treatment. Reports of AEs were obtained through solicited and spontaneous comments from the subjects and through observations by the Investigator as outlined in the study protocol.
Arm/Group | Vehicle Run-In | LME636 | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/213 | 0/69 | 0/65
Serious Adverse Events (participants affected / at risk) | 1/213 | 0/69 | 1/65
Other Adverse Events (participants affected / at risk) | 0/213 | 0/69 | 0/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle Run-In (N=213) | LME636 (N=69) | Vehicle (N=65)
Extradural abscess (Infections and infestations) | 1 | 0 | 0 — The subject who presented extradural abscess discontinued the study due to this AE, which was not related to the investigational product.
Pneumonia (Infections and infestations) | 0 | 0 | 1 — Not related to investigational product

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.